CLINICAL TRIAL: NCT04129190
Title: Single Non-fasting OGTT Versus Fasting OGTT for Screening of Hyperglycaemia in Pregnancy (HIP)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Isra University (Other)
Responsible Party: Principal Investigator, Dr shabeen, Professor, Isra University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IsraU
Record Dates: First submitted 2019-10-15; First posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Diabetes in Pregnancy
MeSH Terms: conditions — Diabetes, Gestational | interventions — Glucose

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single (Experimental)
  Interventions: Biological: Glucose

INTERVENTIONS:
Biological: Glucose — Oral Intake of Glucose

SUMMARY:
With the increasing prevalence of diabetes in pregnancy it is necessary to design a simple, sensitive, cost effective method for screening of hyperglycaemia in pregnancy specially in resource constrained settings.

There is no universally agreed screening and diagnostic criteria to detect hyperglycemia in pregnancy. In present study, DIPSI (non-fasting OGTT) is compared with fasting oral glucose tolerance test (OGTT) to evaluate sensitivity and specificity of both methods in our population.

ELIGIBILITY:
Inclusion Criteria:

All pregnant women

Exclusion Criteria:

Known diabetic

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2019-10-15 (Estimated); Primary Completion 2020-01-15 (Estimated); Study Completion 2020-01-15 (Estimated)

PRIMARY OUTCOMES:
Oral Glucose Tolerance | 2 hours
  Measurement of Plasma Glucose after intake of 75 gram oral glucose

CONTACTS AND LOCATIONS:
Locations (1):
- Isra University, Karachi Campus, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No